CLINICAL TRIAL: NCT00831051
Title: A Double-Blind, Randomized, Multi-Center, Repeat-Dose, Comparison of the Analgesic Efficacy and Safety of the Opioid Combination Q8003 to Each of the Individual Milligram Components (Oxycodone and Morphine) in the Management of Acute Moderate to Severe Pain Following Bunionectomy Surgery
Brief Title: Comparison of the Efficacy and Safety of Q8003 Versus Its Individual Components in Bunionectomy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q8003-021
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: Bunionectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — MoxDuo; Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Q8003 12mg/8mg (Experimental): Combination
  Interventions: Drug: Q8003
- Morphine sulfate 12 mg (Active Comparator): Single component
  Interventions: Drug: Morphine sulfate
- Oxycodone HCl 8mg (Active Comparator): Single component
  Interventions: Drug: Oxycodone HCl
- Q8003 6mg/4mg (Experimental): Combination
  Interventions: Drug: Q8003
- Morphine sulfate 6mg (Active Comparator): Single component
  Interventions: Drug: Morphine sulfate
- Oxycodone HCl 4mg (Active Comparator): Single component
  Interventions: Drug: Oxycodone HCl 4mg

INTERVENTIONS:
Drug: Q8003 — One Q8003 (morphine sulfate and oxycodone HCl) 12mg/8mg IR Capsule q6h
  Arms: Q8003 12mg/8mg
Drug: Morphine sulfate — One morphine sulfate 12mg IR capsule q6h
  Arms: Morphine sulfate 12 mg
Drug: Oxycodone HCl — One oxycodone HCl 8mg IR Capsule q6h
  Arms: Oxycodone HCl 8mg
Drug: Q8003 — One Q8003 (morphine sulfate and oxycodone HCl) 6mg/4mg IR Capsule q6h
  Arms: Q8003 6mg/4mg
Drug: Morphine sulfate — Two morphine sulfate 3mg IR capsules q6h
  Arms: Morphine sulfate 6mg
Drug: Oxycodone HCl 4mg — Two oxycodone HCl 2mg IR Capsules q6h
  Arms: Oxycodone HCl 4mg

SUMMARY:
This is a randomized, double-blind, multicenter, fixed dose factorial study of Q8003 12 mg/8 mg and Q8003 6 mg/4 mg versus its individual morphine sulfate and oxycodone hydrochloride components for the management of acute moderate to severe postoperative pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 18 years of age.
* Females must be non-pregnant, non-lactating, and practicing an acceptable method of birth control, or be surgically sterile or postmenopausal (amenorrhea for ≥ 12 months). Non-pregnancy will be confirmed by pregnancy tests conducted at Screening and Pre-treatment.
* Patient is scheduled for bunionectomy surgery, meets the criteria of an ASA Class I to III, and is willing to stay in the study center for at least 48 hours from the initial dose of study medication post surgery.
* To be randomized after surgery, the patient must report moderate to severe pain (a score of 2 or more on the 4 point Likert scale or at least 4 on the 11 point NPRS scale).

Exclusion Criteria:

* In the opinion of the Investigator, has a history of pulmonary, cardiovascular (including uncontrolled hypertension), neurologic, endocrine, hepatic, gastrointestinal, or kidney disease or therapy that, in the opinion of the Investigator, would jeopardize the patient's well being by participation in this study or is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.
* Used opiates continuously (including tramadol) for more than ten days in the past year.
* Hypersensitivity or poor tolerance to ibuprofen or short term opioids.
* Currently receiving any medications that are not at a stable dose (the same dose for > 2 months prior to date of surgery).
* Was dosed with another investigational drug within 30 days prior to the Screening Visit or has previously received treatment with Q8003.
* Current therapy with central nervous system depressant medications that might increase the risks of treatment with opioids (other than those used with surgical anesthesia).
* Current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Difference in pain intensity scores from baseline | 48 hours

SECONDARY OUTCOMES:
Safety: adverse events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patricia T. Richards, MD, Ph.D., Study Director — QRxPharma Inc.
Locations (6):
- United States (6):
  - Associated Foot and Ankle Specialists, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Crossroads Research, Inc., Owings Mills, Maryland
  - Chesapeake Foot and Ankle, Pasadena, Maryland
  - Advanced Regional Center for Ankle and Foot Care, Altoona, Pennsylvania
  - Jean Brown Research, Salt Lake City, Utah